CLINICAL TRIAL: NCT00530166
Title: A Randomized, Double-Blind, Placebo Controlled, Parallel Group Study to Investigate the Effect of JNJ-18054478 in Subjects With Asthma
Brief Title: Effectiveness and Safety Study for JNJ-18054478 in Asthma Patients.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy following an interim analysis
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR013087; 18054478NAP2002
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Asthma
Keywords: Asthma; persistant asthma; controller medications; FEV1
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 002 (Experimental): sham comparator 3(100 mg) tablets once daily for 12 weeks
  Interventions: Drug: sham comparator
- 001 (Experimental): JNJ-18054478 3(100 mg) tablets once daily for 12 weeks
  Interventions: Drug: JNJ-18054478

INTERVENTIONS:
Drug: JNJ-18054478 — 3(100 mg) tablets once daily for 12 weeks
  Arms: 001
Drug: sham comparator — 3(100 mg) tablets once daily for 12 weeks
  Arms: 002

SUMMARY:
The purpose of this study is to assess the effectiveness of JNJ-18054478 measured by the percent change from baseline in Forced Expiratory Volume in one Second (FEV1) after 12 weeks of therapy in patients with persistent asthma.

DETAILED DESCRIPTION:
Asthma is one of the most common chronic diseases worldwide. This is a randomized (study medication assigned by chance), double-blind study (neither the physician or the patient knows which drug they are receiving, active or placebo) to Investigate the effectiveness and safety of 12 weeks of dosing with JNJ-18054478 (300 mg taken orally once daily) compared with placebo in patients with persistent asthma. The hypothesis is that the study drug will be more effective in treatment of asthma than placebo as measured by the percent change from baseline in Forced Expiratory Volume in one Second (FEV1) after 12 weeks of therapy, without any significant adverse events. Safety evaluations will include, monitoring for adverse reactions, clinical laboratory tests of blood and urine, ECGs to monitor the cardiovascular system, vital signs and physical examinations. Patients will take three capsules (100 mg) of JNJ-18054478 orally once daily for 12 weeks or placebo for the same period.

ELIGIBILITY:
Inclusion Criteria:

* Medically confirmed diagnosis of persistent asthma
* Able to demonstrate reversibility of at least 12% with albuterol inhalation
* Use of short-acting b-2 agonists for rescue >= 5 times within 2 weeks prior
* Able to produce an FEV1 between 45 and 85% of predicted
* Willing to perform study procedures for about 14 weeks.

Exclusion Criteria:

* Use of inhaled corticosteroids within 4 weeks
* Use of oral/parenteral corticosteroids within 8 weeks
* Use of long-acting beta-2 agonists or montelukast within 2 weeks
* History of life-threatening asthma attack within 3 months
* Female of child bearing potential.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-07; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
The percent change from the beginning of the study in Forced Expiratory Volume in one Second (FEV1) after 12 weeks on study drug. | 12 weeks

SECONDARY OUTCOMES:
The change in FEV1 after 1, 2, 4, 6, 8 and 10 weeks therapy. The change in symptoms and use of asthma rescue medication. The number of asthma attacks compared to placebo. The safety, tolerability, and blood and urine levels of JNJ-18054478 | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (36):
- United States (29):
  - Scottsdale, Arizona
  - Long Beach, California
  - Los Angeles, California
  - Paramount, California
  - San Jose, California
  - Colorado Springs, Colorado
  - Pueblo, Colorado
  - Chicago, Illinois
  - Normal, Illinois
  - River Forest, Illinois
  - Baltimore, Maryland
  - Boston, Massachusetts
  - North Dartmouth, Massachusetts
  - Plymouth, Minnesota
  - St Louis, Missouri
  - Skillman, New Jersey
  - North Syracuse, New York
  - Rochester, New York
  - Canton, Ohio
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Lake Oswego, Oregon
  - Medford, Oregon
  - Portland, Oregon
  - Chester, Pennsylvania
  - Philadelphia, Pennsylvania
  - Dallas, Texas
  - Madison, Wisconsin
- San José, Costa Rica
- India (6):
  - Bangalore
  - Chennai
  - Hyderabad
  - Mumbai
  - Mysore
  - Vellore